CLINICAL TRIAL: NCT03416621
Title: Project Q Pilot: Examining Different Treatment Modalities to Maximize Cessation Efforts for Light Smokers
Brief Title: Project Q Pilot: Smoking Cessation for Light Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00089760
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Results first posted 2021-02-24 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Tobacco Use Cessation
Keywords: Light Smoker
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: Cognitive behavioral cessation counseling (Active Comparator): Standard smoking cessation plus support text messages
  Interventions: Behavioral: Cognitive behavioral cessation counseling
- Placebo Comparator: Counseling and placebo drug intervention (Placebo Comparator): enhanced cue exposure treatment (lab-based + interactive SMS texting) + DCS placebo
  Interventions: Behavioral: Cognitive behavioral cessation counseling; Behavioral: Counseling and placebo drug intervention
- Active Comparator: Counseling and active drug intervention (Experimental): enhanced cue exposure treatment (lab-based + interactive SMS texting) + active DCS. In addition to an in-person screening visit, we will conduct three in-person treatment visits and an in-person follow-up visit.
  Interventions: Behavioral: Cognitive behavioral cessation counseling; Drug: Counseling and active drug intervention

INTERVENTIONS:
Behavioral: Cognitive behavioral cessation counseling — Standard smoking cessation plus support text messages
Behavioral: Counseling and placebo drug intervention — Enhanced cue exposure treatment (lab-based + interactive SMS texting) + DCS placebo
  Arms: Placebo Comparator: Counseling and placebo drug intervention
Drug: Counseling and active drug intervention — Enhanced cue exposure treatment (lab-based + interactive SMS texting)+ active DCS. In addition to an in-person, screening visit, we will conduct three in-person treatment visits and an in-person follow-up visit.
  Arms: Active Comparator: Counseling and active drug intervention

SUMMARY:
The purpose of this pilot study is to evaluate the feasibility, acceptability, and preliminary efficacy of an intervention to promote smoking cessation among light smokers.

DETAILED DESCRIPTION:
The three-arm randomized controlled trial compares Arm 1) standard smoking cessation plus support text messages, 2) enhanced cue exposure treatment (lab-based + interactive SMS texting) + D-cycloserine placebo, Arm 3)will include a combination of cognitive behavioral cessation counseling, enhanced cue exposure treatment (lab-based + interactive SMS texting) and a cognitive-enhancing drug - D-cycloserine. In addition to an in-person screening visit, we will conduct three in-person treatment visits and an inperson follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old
* Able to read and understand English or Spanish
* Cognitively able to provide informed consent
* Smoke 1-10 cigs/day on at least 4 days in the past month
* Express a desire to quit smoking in the next 30 days
* Access to a cell phone that can send and receive SMS text messages and take and send pictures

Exclusion Criteria:

* Hypertension with a screening blood pressure over 160/100;
* Hypotension with a screening blood pressure of systolic <90 mm Hg, diastolic <60 mm Hg;
* Participants with a history of hypertension may be allowed to participate in the study if the study physician or physician assistant determines that the condition is stable, controlled by medication, and in no way jeopardizes the individual's safety;
* Coronary heart disease, diagnosed by coronary angiogram;
* History of major heart attack;
* Major cardiac rhythm disorder determined by study MD;
* Chest pain in the last month (unless history, exam, indicate a non-cardiac source);
* Symptomatic cardiac disorder (valvular heart disease, heart murmur, heart failure);
* Diagnosis of severe liver disease or kidney disorder;
* Major gastrointestinal problems or disease (Celiac, Crohn's, Ulcerative Colitis)
* Bleeding ulcers in the past 30 days;
* Current, advanced lung disorder/disease (COPD, emphysema);
* Migraine headaches that occur more frequently than once per week;
* Recent, unexplained fainting spells;
* Problems giving blood samples;
* Diabetes not controlled by diet and exercise alone;
* Current cancer or cancer treatment in the past six months (except basal or squamous cell skin cancer);
* HIV, Hepatitis B, or Hepatitis C;
* History of Tuberculosis or recent positive PPD;
* Other major medical condition;
* Current symptomatic, uncontrolled psychiatric disease;
* Diagnosis of serious mental illness, including bipolar disorder and schizophrenia;
* Suicidal ideation within the past month or lifetime occurrence of attempted suicide;
* Current (within 2 weeks) depression determined by PHQ-9 score > 9 or > 0 on item #9
* Bulimia or anorexia;
* Pregnant or nursing;
* Use (within the past 30 days) of:
* Illegal drugs (or if the urine drug screen is positive for Cocaine, Amphetamine, Opiates, Methamphetamines, PCP, Benzodiazepines, or Barbiturates), unless prescribed for management of acute symptoms (tooth extraction, recent surgery);
* Experimental (investigational) drugs;
* Psychiatric medications including antidepressants (MAOIs, St. John's Wort), lithium, anti-psychotics, or any other medications that are known to affect smoking cessation (e.g. clonidine);
* Wellbutrin, bupropion, Zyban, Chantix, varenicline, nicotine patch, nicotine replacement therapy or any other smoking cessation aid.
* Use of cigars, cigarillos, pipes, Hookah, dissolvable nicotine, snuff, chewing tobacco , or e-cigarettes within the past 30 days;
* Positive result on AUDIT-C;
* Self-report of marijuana use ≥ 4 days per week;
* Significant adverse reaction to D-cycloserine in the past;
* Current or recent (in the past 30 days) participation in another smoking study at our Center or another research facility

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Pollak, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center - Cancer Prevention, Detection and Control, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pollak KI, Oliver JA, Pieper C, Davis JM, Gao X, Noonan D, Kennedy D, Granados I, Fish LJ. Cue-based treatment for light smokers: A proof of concept pilot. Addict Behav. 2021 Mar;114:106717. doi: 10.1016/j.addbeh.2020.106717. Epub 2020 Oct 17. PMID 33109394

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental: Cognitive Behavioral Cessation Counseling | Placebo Comparator: Counseling and Placebo Drug Intervention | Active Comparator: Counseling and Active Drug Intervention
Started | 13 | 12 | 6
Completed | 13 | 11 | 1
Not Completed | 0 | 1 | 5

BASELINE CHARACTERISTICS:
Population: In the comparator standard counseling, one enrolled patient withdrew prior to completing the baseline survey. Three participants in the active comparator arm did not complete the baseline survey.
Groups:
- Experimental: Cue-based Treatment: Enhanced cue exposure treatment (lab-based + interactive SMS texting)
  Cognitive behavioral cessation counseling: Standard smoking cessation plus support text messages
- Comparator: Standard Counseling: Cognitive behavioral cessation counseling: Standard smoking cessation plus support text messages
- Total: Total of all reporting groups
Arm/Group | Experimental: Cue-based Treatment | Comparator: Standard Counseling | Active Comparator: Counseling and Active Drug Intervention | Total
Number analyzed (Participants) | 13 | 11 | 3 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (14.8) | 44.2 (18.4) | 43 (24) | 43.2 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 1 | 19
  Male | 3 | 3 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 11 | 10 | 3 | 24
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 7 | 2 | 17
  White | 3 | 4 | 1 | 8
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1
Education: Some college or college grad [Count of Participants; unit: Participants] | 8 | 9 | 3 | 20
Employment status: Employed [Count of Participants; unit: Participants] | 3 | 5 | 2 | 10
Type of smoker [Count of Participants; unit: Participants]
  Daily | 12 | 11 | 3 | 26
  Intermittent | 1 | 0 | 0 | 1
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 5.8 (2.5) | 6.5 (2.0) | 7 (3.6) | 6.1 (2.2)
Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — Measured by the Fagerstrom Test For Nicotine Dependence (FTND). The FTND has a range of 0-10. The higher the Fagerstrom score, the more intense is the patient's physical dependence on nicotine.
  units on a scale | 2.8 (2.1) | 2.3 (1.7) | 1.7 (2.9) | 2.5 (1.9)
Native Light Smoker [Count of Participants; unit: Participants] — Native light smoker is defined as a participant smoker who has never smoked more than 10 cigarettes per day
  Participants | 7 | 8 | 2 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Completion of at Least 2 Study Visits
Description: Feasibility will be determined by number of participants that complete at least 2 study visits.
Time Frame: Approximately 8 weeks
Population: Only one participant in the "Active Comparator" arm completed the study.
Measure: Count of Participants; unit: Participants
Groups:
- Control: Standard Counseling: Cognitive behavioral cessation counseling: Standard smoking cessation plus support text messages
Arm/Group | Experimental: Cue-based Treatment | Control: Standard Counseling | Active Comparator: Counseling and Active Drug Intervention
Number analyzed (Participants) | 13 | 11 | 1
Participants | 10 | 7 | 1

2. Primary Outcome: Number of Participants Who Rated the Intervention Acceptable
Description: Acceptability will be determined by the number of patients rating the intervention usefulness in the experimental and control arms on a 7-point Likert scale, where 1=extremely useless and 7=extremely useful.
Time Frame: Approximately 8 weeks
Population: The primary outcome was defined as acceptability across the entire sample.
Measure: Count of Participants; unit: Participants
Groups:
- Total: Standard smoking cessation plus support text messages
Arm/Group | Total
Number analyzed (Participants) | 25
Participants | 23

3. Secondary Outcome: Number of Participants With Validated Cessation
Description: Biochemically-validated cessation (absence of salivary cotinine) 1 week post-intervention.
Time Frame: 1 week post-intervention
Population: Only one participant in the "Active Comparator" arm completed the study.
Measure: Count of Participants; unit: Participants
Groups:
- Active Comparator: Counseling and Active Drug Intervention: Enhanced cue exposure treatment (lab-based + interactive SMS texting) + active DCS. In addition to an in-person screening visit, we will conduct three in-person treatment visits and an in-person follow-up visit.
  Cognitive behavioral cessation counseling: Standard smoking cessation plus support text messages Counseling and active drug intervention: Enhanced cue exposure treatment (lab-based + interactive SMS texting)+ active DCS. In addition to an in-person, screening visit, we will conduct three in-person treatment visits and an in-person follow-up visit.
Arm/Group | Experimental: Cue-based Treatment | Control: Standard Counseling | Active Comparator: Counseling and Active Drug Intervention
Number analyzed (Participants) | 13 | 11 | 1
Participants | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Experimental: Cognitive Behavioral Cessation Counseling: Standard smoking cessation plus support text messages Cognitive behavioral cessation counseling: Standard smoking cessation plus support text messages
- Placebo Comparator: Counseling and Placebo Drug Intervention: Enhanced cue exposure treatment (lab-based + interactive SMS texting) + DCS placebo Cognitive behavioral cessation counseling: Standard smoking cessation plus support text messages Counseling and placebo drug intervention: Enhanced cue exposure treatment (lab-based + interactive SMS texting) + DCS placebo
Arm/Group | Experimental: Cognitive Behavioral Cessation Counseling | Placebo Comparator: Counseling and Placebo Drug Intervention | Active Comparator: Counseling and Active Drug Intervention
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/6

LIMITATIONS AND CAVEATS:
Findings are not conclusive due to the pilot nature of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT03416621/ICF_002.pdf
  • Study Protocol and Statistical Analysis Plan (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT03416621/Prot_SAP_003.pdf